CLINICAL TRIAL: NCT03344757
Title: Culturally Adapted Cognitive Behavioral Stress and Self-Management (C-CBSM) Intervention for Prostate Cancer
Brief Title: Health Gatherings - For Your Health After Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Northwestern University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Frank Penedo, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20170656; STU00203197 (Other: Northwestern ID); 1R01CA206456-01A1 (NIH)
Record Dates: First submitted 2017-09-27; First posted 2017-11-17 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Prostate Neoplasm; Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasm, Prostate; Genital Diseases, Male; Prostatic Diseases
Keywords: prostate cancer; localized prostate cancer; spanish; latino; hispanic; stress management
MeSH Terms: conditions — Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Genital Diseases, Male; Prostatic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cultural-Cognitive Behavioral Stress Management (CCBSM) (Experimental): Participants randomized to this arm will receive 10 weekly group-based C-CBSM intervention.
  Interventions: Behavioral: Cultural CBSM
- Cognitive Behavioral Stress Management (CBSM) (Active Comparator): Participants randomized to this arm will receive 10 weekly group-based standard CBSM intervention.
  Interventions: Behavioral: Standard CBSM

INTERVENTIONS:
Behavioral: Cultural CBSM — The Culturally Adapted Cognitive Behavioral Stress Management (C-CBSM) Intervention is a 10 weekly in-person group program. Each session will last about 90 minutes. The meetings will give facts on stress, coping with difficult events, managing anger, social support and stress reactions. Participants will also receive information on how to practice relaxation on their own. The delivery of C-CBSM places a greater emphasis on salient sociocultural determinants of symptom burden and Health Related Quality of Life (HRQoL) in Hispanics (e.g., fatalistic attitudes, family interdependence, perceived discrimination, machismo).
  Arms: Cultural-Cognitive Behavioral Stress Management (CCBSM)
Behavioral: Standard CBSM — The standard Cognitive Behavioral Stress Management (CBSM) Intervention is a 10 weekly in-person group program. Each session will last about 90 minutes. The meetings will give facts on stress, coping with difficult events, managing anger, social support and stress reactions. Participants will also receive information on how to practice relaxation on their own.
  Arms: Cognitive Behavioral Stress Management (CBSM)

SUMMARY:
The purpose of this study is to look at the effects of a 10-week stress management in-person group program. The program will study emotions, stress, and stress management techniques (such as relaxation and coping techniques) on quality of life, distress, depression, and physical health in Spanish- speaking, Hispanic/Latino men diagnosed with Prostate Cancer (PC).

DETAILED DESCRIPTION:
This 5-year study evaluates the effects of a 10-week group-based linguistically translated and culturally adapted cognitive-behavioral stress and self-management (C-CBSM) intervention on symptom burden and health related quality of life (HRQoL) in Hispanic men treated for localized prostate cancer (PC). About 80% PC cases are diagnosed as early disease and have a 5- and 10-year survival rate of almost 100% and 99%, respectively.1 Most patients receive active treatment (~70%) leading to prolonged treatment-related side effects and dysfunction persisting well beyond primary treatment. Survival is offset by chronic side effects such as sexual and urinary dysfunction, pain and fatigue that can lead to poor psychosocial functioning, impaired intimacy and social functioning, and masculinity concerns. Hispanic PC survivors report lower physical and social functioning, poorer emotional well-being and greater sexual and urinary dysfunction, even after accounting for SES and disease severity. These sequelae can lead to elevated glucocorticoid release and inflammatory cytokines that have a direct effect on these symptoms and can interfere with physiological pathways necessary for recovery of sexual and urinary functioning. We have shown that CBSM reduces symptom burden and improves HRQoL in bilingual Hispanic PC survivors. In a pilot we showed that a linguistic translation of CBSM with attention to sociocultural processes improved symptom burden and HRQoL in Spanish monolingual PC survivors. We have also shown that CBSM is associated with reduced glucocorticoid resistance and inflammatory gene expression pathways in circulating leukocytes among breast cancer survivors. We propose to (a) deliver a culturally adapted C-CBSM intervention in Spanish that places greater emphasis on salient sociocultural determinants of symptom burden and HRQoL in Hispanics (e.g., fatalistic attitudes, family interdependence, perceived discrimination, machismo), (b) incorporate a neuroimmune model of symptom regulation and management, and (c) test the efficacy of C-CBSM, relative to standard non-culturally adapted CBSM, in two diverse Hispanic communities (Chicago & Miami). We will test our aims in 200 Hispanic men post-treatment for localized PC with elevated symptom burden in a 2 x 4 randomized design with condition (C-CSBM vs. CBSM) as the between groups factors, and time (baseline, post-intervention & 6- and 12-months post intervention) as the within groups factor.

Our Primary Aim is to determine whether randomization to C-CBSM, relative to standard CBSM, is associated with reduced symptom burden and improved HRQoL. Our Secondary Aims evaluate whether C-CBSM leads to greater improvements in the intervention targets (e.g., stress management, psychological distress & interpersonal disruption), and physiologic adaptation (i.e., glucocorticoid receptor sensitivity & inflammatory gene expression). We will also evaluate psychosocial and physiological mechanisms as mediators of C-CBSM's effects on our primary outcomes. We also explore several moderators (e.g., SES, acculturation, treatment, Hispanic origin) of CCBSM's effect on primary outcomes and the effects of C-CBSM on cardiometabolic health (e.g., lipids, fasting glucose) via reduced inflammation.

Primary Aim:

Aim 1: Determine whether participation in C-CBSM is associated with significantly greater reductions in symptom burden and improvements in HRQoL relative to participation in CBSM.

Secondary Aims:

Aim 2: Determine whether participation in C-CBSM is associated with significantly greater improvements in intervention targets (i.e., improved stress management, and reduced psychological distress and interpersonal disruption) relative to participation in the CBSM condition.

Exploratory Aims:

Aim 3: Explore whether participation in C-CBSM is associated with significantly greater activation of leukocyte glucocorticoid receptor and less inflammatory gene expression profiles relative to CBSM.

Aim 4: Explore whether C-CBSM related improvements in symptom burden and HRQoL are mediated by improvements in intervention targets and gene expression profiles.

Aim 5: Explore moderators of C-CBSM (e.g., SES, treatment type, acculturation, Hispanic ancestry) and CCBSM's effects on cardiometabolic markers via reduced inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age;
2. Hispanic/Latino self-identification;
3. Spanish speakers (including bilinguals who express interest in a Spanish-based psychosocial intervention);
4. Primary diagnosis of localized Prostate Cancer (T1-T3, N0, M0);
5. Surgical or radiation treatment (e.g., external beam, brachytherapy, proton) within minimum of 4 months and maximum of 72-months;
6. Some patients with prior inpatient psychiatric treatment for severe mental illness or overt signs of severe psychopathology (e.g., psychosis) may be enrolled, per P.I. discretion, based on a case-by-case review;
7. Willingness to be randomized and followed for approximately12 months.

Exclusion Criteria:

1. History of non-skin cancer within the last 2 years.
2. Prior inpatient psychiatric treatment for severe mental illness or overt signs of severe psychopathology (e.g., psychosis) within the past six months, as these conditions can interfere with adequate participation in our experimental conditions may be exclusionary, per P.I. discretion, based on a case-by-case review;
3. Active alcohol dependence within the past six months may be exclusionary, per P.I. discretion, based on a case-by-case review;
4. Active substance dependence within the past six months may be exclusionary, per P.I. discretion, based on a case-by-case review; and
5. Acute or chronic immune system medical conditions, medications or conditions that impact immune and endocrine function (e.g., Chronic Fatigue Syndrome (CFS), Lupus, rheumatoid arthritis, Hepatitis C, or immunosuppressive treatment requiring conditions), per PI discretion based on a case by case review.
6. Individuals scoring >3 on the SPMSQ will be excluded or per PI discretion based on a case by case review.

   .

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Penedo, Ph.D., Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pedreira PB, Fleszar-Pavlovic SE, Walsh EA, Noriega Esquives B, Moreno PI, Perdomo D, Heller AS, Antoni MH, Penedo FJ. Familism, family cohesion, and health-related quality of life in Hispanic prostate cancer survivors. J Behav Med. 2024 Aug;47(4):595-608. doi: 10.1007/s10865-024-00479-1. Epub 2024 Mar 1. PMID 38429598

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cultural-Cognitive Behavioral Stress Management (CCBSM) | Cognitive Behavioral Stress Management (CBSM)
Started | 100 | 88
Completed | 82 | 70
Not Completed | 18 | 18
Not completed — Withdrawal by Subject | 18 | 16
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cultural-Cognitive Behavioral Stress Management (CCBSM) | Cognitive Behavioral Stress Management (CBSM) | Total
Number analyzed (Participants) | 100 | 88 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.07 (7.64) | 65.42 (8.42) | 65.77 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 100 | 88 | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 100 | 88 | 188
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 75 | 72 | 147
  More than one race | 15 | 10 | 25
  Unknown or Not Reported | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Symptom Burden as Measure by EPIC-S.
Description: Symptom Burden will be measured using the 5-item sexual domain of the Expanded Prostate Cancer Index Composite (EPIC) - Short Form (EPIC-S). All items are transformed to a 0-100 scale and averaged to calculate the domain summary scores, where higher scores indicate better functioning and less bother.
Time Frame: Baseline, Month 3, Month 6, Month 12
Population: Not all participants completed every assessment/timepoint and some were lost to follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cultural-Cognitive Behavioral Stress Management (CCBSM) | Cognitive Behavioral Stress Management (CBSM)
Number analyzed (Participants) | 100 | 88
score on a scale
  Baseline | 30.1 (2.53) | 32.1 (3.02)
  Month 3: number analyzed (Participants) | 82 | 75
  Month 3 | 34.7 (3.01) | 35.8 (3.30)
  Month 6: number analyzed (Participants) | 69 | 69
  Month 6 | 35.9 (3.39) | 38.0 (3.67)
  Month 12: number analyzed (Participants) | 81 | 70
  Month 12 | 36.2 (3.27) | 38.9 (3.50)

2. Primary Outcome: Change in HRQoL as Measured by the FACT Questionnaire.
Description: HRQoL will be measured using Functional Assessment of Cancer Therapy - Prostate (FACT-P) including 4 domains of the FACT-General (FACT-G). The questionnaire has 39 items, with the total score ranging from 0-156. Higher scores indicate better function.
Time Frame: Baseline, Month 3, Month 6, Month 12
Population: Not all participants completed every assessment/timepoint and some were lost to follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cultural-Cognitive Behavioral Stress Management (CCBSM) | Cognitive Behavioral Stress Management (CBSM)
Number analyzed (Participants) | 100 | 88
score on a scale
  Baseline: number analyzed (Participants) | 99 | 88
  Baseline | 81.1 (1.12) | 81.7 (1.70)
  Month 3: number analyzed (Participants) | 82 | 76
  Month 3 | 83.8 (1.30) | 83.7 (1.45)
  Month 6: number analyzed (Participants) | 71 | 68
  Month 6 | 83.6 (1.51) | 83.3 (1.74)
  Month 12: number analyzed (Participants) | 82 | 70
  Month 12 | 82.6 (1.41) | 83.0 (1.54)

3. Primary Outcome: Change in Symptom Burden as Measure by EPIC-UIN.
Description: Symptom Burden will be measured using the 9-item urinary domain of the Expanded Prostate Cancer Index Composite (EPIC) - Short Form (EPIC-UIN). All items are transformed to a 0-100 scale and averaged to calculate the domain summary scores, where higher scores indicate better functioning and less bother.
Time Frame: Baseline, Month 3, Month 6, Month 12
Population: Not all participants completed every assessment/timepoint and some were lost to follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cultural-Cognitive Behavioral Stress Management (CCBSM) | Cognitive Behavioral Stress Management (CBSM)
Number analyzed (Participants) | 100 | 88
score on a scale
  Baseline | 73.5 (2.45) | 78.8 (2.32)
  Month 3: number analyzed (Participants) | 82 | 75
  Month 3 | 77.4 (2.50) | 82.2 (2.38)
  Month 6: number analyzed (Participants) | 71 | 69
  Month 6 | 79.5 (2.47) | 84.6 (2.18)
  Month 12: number analyzed (Participants) | 82 | 70
  Month 12 | 78.3 (2.41) | 83.3 (2.31)

4. Primary Outcome: Change in HRQoL as Measured by the PROMIS Fatigue Questionnaire
Description: HRQoL will be measured using Patient-Reported Outcome Measurement Information System (PROMIS) short form for Fatigue Questionnaire. The PROMIS Fatigue measure generates t-scores with a mean of 50 and a standard deviation of 10. Scores typically range from approximately 30 to 80. Higher scores indicate greater fatigue.
Time Frame: Baseline, Month 3, Month 6, Month 12
Population: Not all participants completed every assessment/timepoint and some were lost to follow-up.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Cultural-Cognitive Behavioral Stress Management (CCBSM) | Cognitive Behavioral Stress Management (CBSM)
Number analyzed (Participants) | 100 | 88
T-score
  Baseline | 43.2 (0.90) | 43.5 (0.99)
  Month 3: number analyzed (Participants) | 82 | 75
  Month 3 | 43.3 (0.88) | 42.8 (1.06)
  Month 6: number analyzed (Participants) | 70 | 69
  Month 6 | 43.9 (1.09) | 43.1 (1.05)
  Month 12: number analyzed (Participants) | 82 | 70
  Month 12 | 43.5 (0.96) | 43.0 (0.99)

5. Primary Outcome: Change in HRQoL as Measured by the PROMIS Pain Questionnaire
Description: HRQoL will be measured using the PROMIS short form for Pain Interference Questionnaire. The items are item banks, and scoring is done via a computer adaptive test (CAT), which utilizes item response theory (IRT) to calculate a score that is then transformed into a T-score with a mean of 50 and a standard deviation of 10. Scores typically range from approximately 30 to 80. Items are administered in an iterative approach where subsequent items are calibrated on prior ones. Once standard error reaches 2 or less, the CAT stops administering items. Higher scores indicate greater pain interference.
Time Frame: Baseline, Month 3, Month 6, Month 12
Population: Not all participants completed every assessment/timepoint and some were lost to follow-up.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Cultural-Cognitive Behavioral Stress Management (CCBSM) | Cognitive Behavioral Stress Management (CBSM)
Number analyzed (Participants) | 100 | 88
T-score
  Baseline | 47.8 (0.93) | 47.0 (0.97)
  Month 3: number analyzed (Participants) | 82 | 75
  Month 3 | 46.7 (0.96) | 46.4 (1.08)
  Month 6: number analyzed (Participants) | 70 | 69
  Month 6 | 47.1 (1.20) | 46.9 (1.06)
  Month 12: number analyzed (Participants) | 82 | 70
  Month 12 | 48.3 (1.07) | 46.2 (1.02)

6. Secondary Outcome: Change in Stress Management Skills as Measured by MOCS-A
Description: Stress management skills will be measured using the Measure of Current Status Part A (MOCS-A) Questionnaire. MOCS-A is a 13-item questionnaire with a total score ranging from 0 - 52 with the higher score indicating greater stress management skills.
Time Frame: Baseline, Month 3, Month 6, Month 12
Population: Not all participants completed every assessment/timepoint and some were lost to follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cultural-Cognitive Behavioral Stress Management (CCBSM) | Cognitive Behavioral Stress Management (CBSM)
Number analyzed (Participants) | 100 | 88
score on a scale
  Baseline: number analyzed (Participants) | 99 | 88
  Baseline | 38.5 (0.87) | 37.6 (1.09)
  Month 3: number analyzed (Participants) | 82 | 74
  Month 3 | 38.6 (0.91) | 38.3 (1.09)
  Month 6: number analyzed (Participants) | 70 | 69
  Month 6 | 39.6 (0.93) | 39.3 (1.23)
  Month 12: number analyzed (Participants) | 81 | 70
  Month 12 | 39.2 (0.90) | 38.0 (0.95)

7. Secondary Outcome: Change in Prostate Cancer-specific Psychological Distress as Measured by MAX-PC - Section I-II
Description: Psychological distress will be measured using the Memorial Anxiety Scale for Prostate Cancer Patients (MAX-PC) Questionnaire. The MAX-PC sections I-II is a 14-item questionnaire with a total score ranging from 0-42 with the higher score indicating increased distress.
Time Frame: Baseline, Month 3, Month 6, Month 12
Population: Not all participants completed every assessment/timepoint and some were lost to follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cultural-Cognitive Behavioral Stress Management (CCBSM) | Cognitive Behavioral Stress Management (CBSM)
Number analyzed (Participants) | 100 | 88
score on a scale
  Baseline | 7.1 (0.94) | 10.0 (1.20)
  Month 3: number analyzed (Participants) | 82 | 75
  Month 3 | 5.6 (0.98) | 6.2 (0.97)
  Month 6: number analyzed (Participants) | 71 | 67
  Month 6 | 5.01 (0.93) | 7.7 (1.24)
  Month 12: number analyzed (Participants) | 82 | 70
  Month 12 | 6.7 (1.08) | 6.1 (0.94)

8. Secondary Outcome: Change in Prostate Cancer-specific Psychological Distress as Measured by MAX-PC - Section III
Description: Psychological distress will be measured using the Memorial Anxiety Scale for Prostate Cancer Patients (MAX-PC) Questionnaire. The MAX-PC section III is a 4-item questionnaire with a total score ranging from 0-12 with the lower score indicating increased distress.
Time Frame: Baseline, Month 3, Month 6, Month 12
Population: Not all participants completed every assessment/timepoint and some were lost to follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cultural-Cognitive Behavioral Stress Management (CCBSM) | Cognitive Behavioral Stress Management (CBSM)
Number analyzed (Participants) | 100 | 88
score on a scale
  Baseline | 8.5 (0.28) | 8.1 (0.37)
  Month 3: number analyzed (Participants) | 82 | 75
  Month 3 | 8.9 (0.31) | 9.1 (0.33)
  Month 6: number analyzed (Participants) | 71 | 67
  Month 6 | 8.7 (0.29) | 8.3 (0.38)
  Month 12: number analyzed (Participants) | 82 | 70
  Month 12 | 9.1 (0.30) | 8.8 (0.35)

9. Secondary Outcome: Change in Psychosocial Distress as Measured by the PROMIS Depression Questionnaire
Description: PROMIS-Depression is a 28-item questionnaire with a total score ranging from 28-140 with the higher score indicating increased symptoms of depression.
Time Frame: Baseline, Month 3, Month 6, Month 12
Population: Not all participants completed every assessment/timepoint and some were lost to follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cultural-Cognitive Behavioral Stress Management (CCBSM) | Cognitive Behavioral Stress Management (CBSM)
Number analyzed (Participants) | 100 | 88
score on a scale
  Baseline | 44.8 (0.91) | 45.9 (0.96)
  Month 3: number analyzed (Participants) | 82 | 75
  Month 3 | 43.8 (0.94) | 44.7 (1.05)
  Month 6: number analyzed (Participants) | 70 | 69
  Month 6 | 44.8 (1.05) | 45.4 (1.12)
  Month 12: number analyzed (Participants) | 82 | 70
  Month 12 | 45.5 (0.97) | 44.9 (1.10)

10. Secondary Outcome: Change in Psychosocial Distress as Measured by the PROMIS Anxiety Questionnaire
Description: PROMIS-Anxiety is a 29-item questionnaire with a total score ranging from 29-145 with the higher score indicating increased symptoms of anxiety.
Time Frame: Baseline, Month 3, Month 6, Month 12
Population: Not all participants completed every assessment/timepoint and some were lost to follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cultural-Cognitive Behavioral Stress Management (CCBSM) | Cognitive Behavioral Stress Management (CBSM)
Number analyzed (Participants) | 100 | 88
score on a scale
  Baseline: number analyzed (Participants) | 100 | 87
  Baseline | 49.5 (0.98) | 50.0 (1.08)
  Month 3: number analyzed (Participants) | 82 | 75
  Month 3 | 50.4 (0.96) | 49.1 (1.18)
  Month 6: number analyzed (Participants) | 70 | 69
  Month 6 | 51.0 (1.16) | 49.8 (1.24)
  Month 12: number analyzed (Participants) | 82 | 70
  Month 12 | 50.7 (0.98) | 49.0 (1.15)

11. Secondary Outcome: Change in Interpersonal Function as Measured the SIP Questionnaire
Description: Sickness Impact Profile (SIP) is a 20-item questionnaire responded with a yes or no. The total number of yes responses will be scored as 1 point with the total score ranging from 0-20 with the higher score indicating poor interpersonal function.
Time Frame: Baseline, Month 3, Month 6, Month 12
Population: Not all participants completed every assessment/timepoint and some were lost to follow-up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cultural-Cognitive Behavioral Stress Management (CCBSM) | Cognitive Behavioral Stress Management (CBSM)
Number analyzed (Participants) | 100 | 88
score on a scale
  Baseline: number analyzed (Participants) | 99 | 87
  Baseline | 2.5 (0.28) | 3.1 (0.38)
  Month 3: number analyzed (Participants) | 80 | 74
  Month 3 | 2.6 (0.40) | 2.9 (0.45)
  Month 6: number analyzed (Participants) | 68 | 64
  Month 6 | 2.2 (0.30) | 2.5 (0.40)
  Month 12: number analyzed (Participants) | 74 | 67
  Month 12 | 2.6 (0.38) | 2.3 (0.36)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Grade 1 Mild; asymptomatic/mild symptoms; clinical or diagnostic observations only; intervention not indicated Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL Grade 4 Life-threatening consequences; urgent intervention indicated Grade 5 Death related to AE
Arm/Group | Cultural-Cognitive Behavioral Stress Management (CCBSM) | Cognitive Behavioral Stress Management (CBSM)
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/88
Serious Adverse Events (participants affected / at risk) | 0/100 | 3/88
Other Adverse Events (participants affected / at risk) | 3/100 | 7/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cultural-Cognitive Behavioral Stress Management (CCBSM) (N=100) | Cognitive Behavioral Stress Management (CBSM) (N=88)
Injury (Injury, poisoning and procedural complications) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Hypertension (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cultural-Cognitive Behavioral Stress Management (CCBSM) (N=100) | Cognitive Behavioral Stress Management (CBSM) (N=88)
COVID-19 (Infections and infestations) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT03344757/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT03344757/ICF_001.pdf